CLINICAL TRIAL: NCT03361748
Title: A Phase 2, Multicenter Study to Determine the Efficacy and Safety of bb2121 in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: Efficacy and Safety Study of bb2121 in Subjects With Relapsed and Refractory Multiple Myeloma
Acronym: KarMMa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB2121-MM-001; U1111-1202-5554 (Other: WHO); 2017-002245-29 (EudraCT Number)
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Efficacy and Safety; BB2121; CAR T Cell; BCMA; Relapsed and Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — idecabtagene vicleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of bb2121 (Experimental): bb2121 autologous CAR T cells will be infused at a dose ranging from 15 - 450 x 10^6 CAR+ T cells after receiving lymphodepleting chemotherapy.
  Interventions: Biological: bb2121

INTERVENTIONS:
Biological: bb2121 — : bb2121 consists of autologous T lymphocytes transduced with an anti-BCMA02 CAR lentiviral vector to express a chimeric antigen receptor targeting the human B cell maturation antigen (anti-BCMA CAR).

SUMMARY:
This is an open label, single-arm, multicenter, Phase 2 study to evaluate the efficacy and safety of bb2121 in subjects with relapsed and refractory multiple myeloma. A leukapheresis procedure will be performed to manufacture bb2121 chimeric antigen receptor (CAR) modified T cells. Prior to bb2121 infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide.

DETAILED DESCRIPTION:
Anti-myeloma bridging treatment is allowed for disease control while bb2121 is being manufactured.

ELIGIBILITY:
Inclusion Criteria:

Eligibility is determined prior to leukapheresis. Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Documented diagnosis of multiple myeloma

   * Must have received at least 3 prior MM treatment regimens. Note: induction with or without hematopoietic stem cell transplant and with or without maintenance therapy is considered a single regimen.
   * Must have undergone at least 2 consecutive cycles of treatment for each regimen, unless PD was the best response to the regimen.
   * Must have received a proteasome inhibitor, an immunomodulatory agent and an anti-CD38 antibody.
   * Must be refractory to the last treatment regimen.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Subjects must have measurable disease, including at least one of the criteria below:

   * Serum M-protein greater or equal to 1.0 g/dL
   * Urine M-protein greater or equal to 200 mg/24 h
   * Serum free light chain (FLC) assay: involved FLC level greater or equal to 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal
5. Recovery to Grade 1 or baseline of any non-hematologic toxicities due to prior treatments, excluding alopecia and Grade 2 neuropathy.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subjects with known central nervous system involvement with myeloma.
2. History or presence of clinically relevant central nervous system (CNS) pathology.
3. Subjects with active or history of plasma cell leukemia.
4. Subjects with solitary plasmacytomas or non-secretory myeloma without other evidence of measurable disease
5. Inadequate organ function
6. Ongoing treatment with chronic immunosuppressants
7. Previous history of an allogeneic hematopoietic stem cell transplantation or treatment with any gene therapy-based therapeutic for cancer or investigational cellular therapy for cancer or BCMA targeted therapy
8. Evidence of human immunodeficiency virus (HIV) infection.
9. Seropositive for and with evidence of active viral infection with hepatitis B virus (HBV)
10. Seropositive for and with evidence of active viral infection with hepatitis B virus (HBV) and Hepatitis C virus (HCV)
11. Subjects with a history of class III or IV congestive heart failure (CHF) or severe non-ischemic cardiomyopathy, history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months.
12. Subjects with second malignancies in addition to myeloma if the second malignancy has required therapy in the last 3 years or is not in complete remission
13. Pregnant or lactating women.
14. Subject with known hypersensitivity to any component of bb2121 productThe presence of any of the following will exclude a subject from enrollment:

1. Subjects with known central nervous system involvement with myeloma. 2. History or presence of clinically relevant central nervous system (CNS) pathology.

3. Subjects with active or history of plasma cell leukemia. 4. Subjects with solitary plasmacytomas or non-secretory myeloma without other evidence of measurable disease 5. Inadequate organ function 6. Ongoing treatment with chronic immunosuppressants 7. Previous history of an allogeneic hematopoietic stem cell transplantation or treatment with any gene therapy-based therapeutic for cancer or investigational cellular therapy for cancer or BCMA targeted therapy 8. Evidence of human immunodeficiency virus (HIV) infection. 9. Seropositive for and with evidence of active viral infection with hepatitis B virus (HBV) and Hepatitis C virus (HCV) 10. Subjects with a history of class III or IV congestive heart failure (CHF) or severe non-ischemic cardiomyopathy, history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months. 11. Subjects with second malignancies in addition to myeloma if the second malignancy has required therapy in the last 3 years or is not in complete remission 12. Pregnant or lactating women. 13 Subject with known hypersensitivity to any component of bb2121 product, cyclophosphamide, fludarabine, or tocilizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb; Kristen Hege, Study Director — Celgene
Locations (48):
- United States (18):
  - Local Institution - 108, San Francisco, California
  - University of California - San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Local Institution - 103, Atlanta, Georgia
  - Local Institution - 107, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Local Institution - 106, Boston, Massachusetts
  - Local Institution - 105, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Local Institution - 102, Hackensack, New Jersey
  - Local Institution - 109, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Local Institution - 101, Nashville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Local Institution - 104, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven, Leuven, Flemish Brabant
  - Local Institution - 201, Leuven
- Canada (2):
  - Local Institution - 301, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto
- France (4):
  - Centre Hospitalier Regional Universitaire de Lille-Hopital Calude Huriez Service des Maladies du Sang, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Nantes - Hotel Dieu, Nantes, Pays de la Loire Region
  - Local Institution - 402, Lille
  - Local Institution - 401, Nantes
- Germany (6):
  - Universitatsklinikum Heidelberg Medizinische Klinik Krehl-Klinik Haematologie, Onkologie, Rheumato, Heidelberg, Baden-Wurttemberg
  - University of Tübingen, Tübingen, Baden-Wurttemberg
  - Universitatsklinikum Würzburg, Würzburg, Bavaria
  - Local Institution - 502, Heidelberg
  - Local Institution - 503, Tübingen
  - Local Institution - 501, Würzburg
- Italy (4):
  - Azienda Ospedaliero Universitaria Di Bologna Policlinico, Bologna, Emilia-Romagna
  - Local Institution - 602, Bergamo
  - Ospedali Riuniti di Bergamo, Bergamo
  - Local Institution - 601, Bologna
- Japan (8):
  - Tokai University Hospital, Isehara, Kanagawa
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Japan Red Cross Medical Center, Shibuya-ku, Tokyo
  - Local Institution - 803, Isehara City, Kanagawa
  - Local Institution - 801, Shibuya-ku
  - Local Institution - 802, Shimotsuke
  - Local Institution - 804, Shinjuku
  - Tokyo Women's Medical University Hospital, Shinjuku
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol Can Ruti, Badalona, Barcelona
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Local Institution - 702, Badalona (Barcelona)
  - Local Institution - 701, Pamplona

REFERENCES:
- [Background] Raje N, Berdeja J, Lin Y, Siegel D, Jagannath S, Madduri D, Liedtke M, Rosenblatt J, Maus MV, Turka A, Lam LP, Morgan RA, Friedman K, Massaro M, Wang J, Russotti G, Yang Z, Campbell T, Hege K, Petrocca F, Quigley MT, Munshi N, Kochenderfer JN. Anti-BCMA CAR T-Cell Therapy bb2121 in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2019 May 2;380(18):1726-1737. doi: 10.1056/NEJMoa1817226. PMID 31042825
- [Background] Munshi NC, Anderson LD Jr, Shah N, Madduri D, Berdeja J, Lonial S, Raje N, Lin Y, Siegel D, Oriol A, Moreau P, Yakoub-Agha I, Delforge M, Cavo M, Einsele H, Goldschmidt H, Weisel K, Rambaldi A, Reece D, Petrocca F, Massaro M, Connarn JN, Kaiser S, Patel P, Huang L, Campbell TB, Hege K, San-Miguel J. Idecabtagene Vicleucel in Relapsed and Refractory Multiple Myeloma. N Engl J Med. 2021 Feb 25;384(8):705-716. doi: 10.1056/NEJMoa2024850. PMID 33626253
- [Derived] Sidana S, Ahmed N, Akhtar OS, Brazauskas R, Oloyede T, Bye M, Hansen D, Ferreri C, Freeman CL, Afrough A, Anderson LD Jr, Dhakal B, Dhanda D, Gowda L, Hashmi H, Harrison MJ, Kitali A, Landau H, Mirza AS, Patwardhan P, Qazilbash M, Usmani S, Patel K, Nishihori T, Ganguly S, Pasquini MC. Standard-of-care idecabtagene vicleucel for relapsed/refractory multiple myeloma. Blood. 2025 Jul 10;146(2):167-177. doi: 10.1182/blood.2024026216. PMID 40198886
- [Derived] Delforge M, Otero PR, Shah N, Moshkovich O, Braverman J, Dhanda DS, Lanar S, Devlen J, Miera M, Gerould H, Campbell TB, Munshi NC. Analysis of patient-reported experiences up to 2 years after receiving idecabtagene vicleucel (ide-cel, bb2121) for relapsed or refractory multiple myeloma: Longitudinal findings from the phase 2 KarMMa trial. Leuk Res. 2023 Jun;129:107074. doi: 10.1016/j.leukres.2023.107074. Epub 2023 Apr 3. PMID 37087950
- [Derived] Connarn JN, Witjes H, van Zutphen-van Geffen M, de Greef R, Campbell TB, Hege K, Zhou S, Lamba M. Characterizing the exposure-response relationship of idecabtagene vicleucel in patients with relapsed/refractory multiple myeloma. CPT Pharmacometrics Syst Pharmacol. 2023 Nov;12(11):1687-1697. doi: 10.1002/psp4.12922. Epub 2023 Feb 15. PMID 36794354
- [Derived] Karampampa K, Zhang W, Venkatachalam M, Cotte FE, Dhanda D. Cost-effectiveness of idecabtagene vicleucel compared with conventional care in triple-class exposed relapsed/refractory multiple myeloma patients in Canada and France. J Med Econ. 2023 Jan-Dec;26(1):243-253. doi: 10.1080/13696998.2023.2173466. PMID 36705644
- [Derived] Shah N, Mojebi A, Ayers D, Cope S, Dhanasiri S, Davies FE, Hari P, Patel P, Hege K, Dhanda D. Indirect treatment comparison of idecabtagene vicleucel versus conventional care in triple-class exposed multiple myeloma. J Comp Eff Res. 2022 Jul;11(10):737-749. doi: 10.2217/cer-2022-0045. Epub 2022 Apr 29. PMID 35485211
- [Derived] Sharma P, Kanapuru B, George B, Lin X, Xu Z, Bryan WW, Pazdur R, Theoret MR. FDA Approval Summary: Idecabtagene Vicleucel for Relapsed or Refractory Multiple Myeloma. Clin Cancer Res. 2022 May 2;28(9):1759-1764. doi: 10.1158/1078-0432.CCR-21-3803. PMID 35046063
- [Derived] Delforge M, Shah N, Miguel JSF, Braverman J, Dhanda DS, Shi L, Guo S, Yu P, Liao W, Campbell TB, Munshi NC. Health-related quality of life with idecabtagene vicleucel in relapsed and refractory multiple myeloma. Blood Adv. 2022 Feb 22;6(4):1309-1318. doi: 10.1182/bloodadvances.2021005913. PMID 34933328
- [Derived] Da Via MC, Dietrich O, Truger M, Arampatzi P, Duell J, Heidemeier A, Zhou X, Danhof S, Kraus S, Chatterjee M, Meggendorfer M, Twardziok S, Goebeler ME, Topp MS, Hudecek M, Prommersberger S, Hege K, Kaiser S, Fuhr V, Weinhold N, Rosenwald A, Erhard F, Haferlach C, Einsele H, Kortum KM, Saliba AE, Rasche L. Homozygous BCMA gene deletion in response to anti-BCMA CAR T cells in a patient with multiple myeloma. Nat Med. 2021 Apr;27(4):616-619. doi: 10.1038/s41591-021-01245-5. Epub 2021 Feb 22. PMID 33619368
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 137 participants treated
Groups:
- BB2121: BB2121
Period: Overall Study
Arm/Group | BB2121
Started | 137
Completed (completed as per protocol) | 36
Not Completed | 101
Not completed — Death | 77
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 20

BASELINE CHARACTERISTICS:
Arm/Group | BB2121
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 112
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 103
  More than one race | 0
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Number of participants who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by an independent response committee (IRC).
Time Frame: From first dose to 24 Months
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BB2121
Number analyzed (Participants) | 137
Percentage of Participants | 74.5 [67.1 to 81.8]

2. Secondary Outcome: Complete Response Rate
Description: Percentage of participants who achieved CR or sCR according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by an IRC.
Time Frame: From first dose to 24 Months
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BB2121
Number analyzed (Participants) | 137
Percentage of participants | 34.3 [26.4 to 42.3]

3. Secondary Outcome: Time to Response
Description: Time from first bb2121 infusion to first documentation of response of PR or better.
Time Frame: From first dose to initial response (approximately on average 1.2 months, max of 8.8 months)
Population: All Treated Participants with a CR or PR as per IRC
Measure: Median (Full Range); unit: Months
Arm/Group | BB2121
Number analyzed (Participants) | 102
Months | 1.0 [0.5 to 8.8]

4. Secondary Outcome: Duration of Response
Description: Time from first documentation of response or PR or better to first documentation of disease progression or death from any cause, whichever occurs first.
Time Frame: From first dose to 24 months after first dose
Population: All Treated Participants with a CR or PR as per IRC
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BB2121
Number analyzed (Participants) | 102
Months | 11.04 [9.92 to 12.52]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from first bb2121 infusion to first documentation of progressive disease (PD), or death due to any cause, whichever occurs first.
Time Frame: From first dose to 24 months after first dose
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BB2121
Number analyzed (Participants) | 137
Months | 8.90 [6.01 to 11.86]

6. Secondary Outcome: Time to Progression (TTP)
Description: as for outcome 5
Time Frame: From first dose to 24 months after first dose
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BB2121
Number analyzed (Participants) | 137
Months | 10.38 [6.11 to 12.06]

7. Secondary Outcome: Overall Survival
Description: Time from first bb2121 infusion to time of death due to any cause.
Time Frame: From screening to the end of follow up (approximately 5 years and 2 months)
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BB2121
Number analyzed (Participants) | 137
Months | 28.25 [20.21 to 38.08]

8. Secondary Outcome: Number of Participants With Safety Related Events
Description: Number of participants with adverse events (AEs), adverse events of special interest (AESI), serious adverse events (SAEs), cytokine release syndrome, neurotoxicity, infection and clinically signifcant laboratory abnormalities.
Time Frame: From screening to the end of follow up (approximately 5 years and 2 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | BB2121
Number analyzed (Participants) | 137
Participants
  Any Grade AE | 137
  Grade 3 or 4 AE | 136
  SAEs | 98
  AEs of Special Interest | 136
  Cytokine Release Syndrome | 116
  Neurotoxicity | 53
  Infections | 95
  Clinically Significant Laboratory Abnormalities | 0

9. Secondary Outcome: Cmax
Description: Cmax is defined as the maximum transgene level at Tmax
  Tmax: The time of maximum observed transgene level, obtained directly from the observed transgene level - time.
Time Frame: From first dose to the end of follow up (Approximately 5 years)
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: transgene copies/ug of genomic DNA
Arm/Group | BB2121
Number analyzed (Participants) | 136
transgene copies/ug of genomic DNA
  Total | 388150.65 (372280.64)
  450x10^6 cells: number analyzed (Participants) | 63
  450x10^6 cells | 449826.92 (375293.18)
  300x10^6 cells: number analyzed (Participants) | 69
  300x10^6 cells | 335916.20 (369546.39)
  150x10^6 cells: number analyzed (Participants) | 4
  150x10^6 cells | 317793.50 (284926.30)

10. Secondary Outcome: AUC 0-9M
Description: The AUC of the transgene level from the time of dosing to 9 months
Time Frame: at 9 months post first dose (Approximtately 9 Months)
Population: PK Evaluable Population for AUC at 9 Months
Measure: Mean (Standard Deviation); unit: copies*days/ug
Arm/Group | BB2121
Number analyzed (Participants) | 122
copies*days/ug
  Total | 8634034.70 (9909488.82)
  450x10^6 cells: number analyzed (Participants) | 60
  450x10^6 cells | 10599751.18 (10833877.42)
  300x10^6 cells: number analyzed (Participants) | 60
  300x10^6 cells | 6604279.35 (8523928.48)
  150x10^6 cells: number analyzed (Participants) | 2
  150x10^6 cells | 10555200.59 (13555457.13)

11. Secondary Outcome: Tmax
Description: Tmax: The time of maximum observed transgene level, obtained directly from the observed transgene level - time.
Time Frame: From first dose to the end of follow up (Approximately 5 years)
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | BB2121
Number analyzed (Participants) | 136
Days
  Total | 12.07 (4.114)
  450x10^6 cells: number analyzed (Participants) | 63
  450x10^6 cells | 12.37 (4.513)
  300x10^6 cells: number analyzed (Participants) | 69
  300x10^6 cells | 11.74 (3.830)
  150x10^6 cells: number analyzed (Participants) | 4
  150x10^6 cells | 13.25 (1.500)

12. Secondary Outcome: Number of Participants With Anti-CAR-Antibodies
Description: Number of Participants with Anti-CAR-Antibodies.
  Pre-postive is defined by last value before or on bb2121 infusion date is positive Post-positve is defined by at least one positive value post bb2121 infusion.
Time Frame: From first dose to the end of follow up (Approximately 5 years)
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | BB2121
Number analyzed (Participants) | 137
Participants
  Pre-Positive Pre-positive and post-positive: number analyzed (Participants) | 6
  Pre-Positive Pre-positive and post-positive | 6
  Pre-Positive Pre-positive and post-negative: number analyzed (Participants) | 6
  Pre-Positive Pre-positive and post-negative | 0
  Pre-Positive Missing post data: number analyzed (Participants) | 6
  Pre-Positive Missing post data | 0
  Pre-Negative Pre-negative and post-postive: number analyzed (Participants) | 130
  Pre-Negative Pre-negative and post-postive | 69
  Pre-Negative Pre-negative and post-negative: number analyzed (Participants) | 130
  Pre-Negative Pre-negative and post-negative | 60
  Pre-Negative Missing post data: number analyzed (Participants) | 130
  Pre-Negative Missing post data | 1
  Missing Pre Data Post-positive: number analyzed (Participants) | 1
  Missing Pre Data Post-positive | 1
  Missing Pre Data post-negative: number analyzed (Participants) | 1
  Missing Pre Data post-negative | 0
  Missing Pre Data missing Post Data: number analyzed (Participants) | 1
  Missing Pre Data missing Post Data | 0

13. Secondary Outcome: Percentage of Participants Who Achieved >= VGPR and MRD Negative Status
Description: Percentage of participants who achieved ≥ VGPR and MRD negative status at a sensitivity of 10-⁵ at any time point within 3 months prior to achieving at least VGPR until the time of PD/death.
  MRD in the bone marrow will be measured using both next generation sequencing (NGS) techniques measuring immunoglobulin gene rearrangements of the malignant clone.
  MRD will be reported with a sensitivity of 10-⁴, 10-⁵, and 10-⁶ nucleated cells. The primary analysis for MRD negative response will use the sensitivity of 10-⁵.
  MRD = Minimal Residual Disease PD = Progressive Disease VGPR = Very good partial response.
Time Frame: From screening to the end of follow up (Approximately 5 years and 2 months)
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BB2121
Number analyzed (Participants) | 137
Percentage of Participants
  10^(-4) Sensitivity | 41.6 [33.3 to 50.3]
  10^(-5) Sensitivity | 40.9 [32.6 to 49.6]
  10^(-6) Sensitivity | 24.8 [17.8 to 32.9]

14. Secondary Outcome: Mean Change From Baseline on the EORTC QLQ-C30 - Fatigue.
Description: Mean change from baseline on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
  The QLQ-C30 employs a week recall period for all items. All items will be scored from 0 to 100. The average of the scores will represent the symptoms score. A high score for a symptom scale/item represents a high level of symptomatic problem.
Time Frame: At Day 1 and at specific time points up to month 24
Population: PRO Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BB2121
Number analyzed (Participants) | 126
Score on a Scale
  Day 1: number analyzed (Participants) | 114
  Day 1 | 4.4 (18.56)
  Month 1: number analyzed (Participants) | 109
  Month 1 | 1.1 (24.38)
  Month 3: number analyzed (Participants) | 86
  Month 3 | -10.1 (24.32)
  Month 6: number analyzed (Participants) | 76
  Month 6 | -15.1 (24.39)
  Month 9: number analyzed (Participants) | 59
  Month 9 | -21.5 (24.58)
  Month 12: number analyzed (Participants) | 55
  Month 12 | -16.4 (25.02)
  Month 18: number analyzed (Participants) | 26
  Month 18 | -18.4 (19.10)
  Month 24: number analyzed (Participants) | 14
  Month 24 | -7.9 (15.97)

15. Secondary Outcome: Mean Change From Baseline on the EORTC QLQ-C30 - Pain
Description: as for outcome 14
Time Frame: At Day 1 and at specific time points up to month 24
Population: PRO Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BB2121
Number analyzed (Participants) | 126
Score on a Scale
  Day 1: number analyzed (Participants) | 114
  Day 1 | -3.8 (19.46)
  Month 1: number analyzed (Participants) | 109
  Month 1 | -8.9 (26.02)
  Month 3: number analyzed (Participants) | 86
  Month 3 | -12.0 (26.65)
  Month 6: number analyzed (Participants) | 76
  Month 6 | -14.5 (26.15)
  Month 9: number analyzed (Participants) | 59
  Month 9 | -17.5 (24.26)
  Month 12: number analyzed (Participants) | 55
  Month 12 | -17.3 (26.05)
  Month 18: number analyzed (Participants) | 26
  Month 18 | -16.7 (25.39)
  Month 24: number analyzed (Participants) | 14
  Month 24 | -13.1 (16.25)

16. Secondary Outcome: Mean Change From Baseline on the EORTC QLQ-C30 - Physical Functioning
Description: The QLQ-C30 employs a week recall period for all items. All items will be scored from 0 to 100 and an average will be taken. This average is the overall score. A higher scale score represents a higher level of well-being and better ability of daily functioning. Thus, a high score for a functional scale represents a high/healthy level of functioning.
Time Frame: At Day 1 and at specific time points up to month 24
Population: PRO Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BB2121
Number analyzed (Participants) | 126
Score on a Scale
  Day 1: number analyzed (Participants) | 114
  Day 1 | -0.4 (18.13)
  Month 1: number analyzed (Participants) | 109
  Month 1 | 2.1 (22.27)
  Month 3: number analyzed (Participants) | 86
  Month 3 | 9.8 (18.54)
  Month 6: number analyzed (Participants) | 76
  Month 6 | 13.9 (18.47)
  Month 9: number analyzed (Participants) | 59
  Month 9 | 13.1 (19.02)
  Month 12: number analyzed (Participants) | 55
  Month 12 | 13.3 (19.16)
  Month 18: number analyzed (Participants) | 26
  Month 18 | 12.8 (15.99)
  Month 24: number analyzed (Participants) | 14
  Month 24 | 3.8 (13.77)

17. Secondary Outcome: Mean Change From Baseline on the EORTC QLQ-C30 - Cognitive Functioning
Description: as for outcome 16
Time Frame: At Day 1 and at specific time points up to month 24
Population: PRO Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BB2121
Number analyzed (Participants) | 126
Score on a Scale
  Day 1: number analyzed (Participants) | 114
  Day 1 | -0.4 (16.66)
  Month 1: number analyzed (Participants) | 109
  Month 1 | 2.8 (20.10)
  Month 3: number analyzed (Participants) | 86
  Month 3 | 5.4 (17.42)
  Month 6: number analyzed (Participants) | 76
  Month 6 | 6.4 (16.55)
  Month 9: number analyzed (Participants) | 59
  Month 9 | 6.8 (14.88)
  Month 12: number analyzed (Participants) | 55
  Month 12 | 4.2 (17.63)
  Month 18: number analyzed (Participants) | 26
  Month 18 | 3.8 (19.61)
  Month 24: number analyzed (Participants) | 14
  Month 24 | 3.6 (16.25)

18. Secondary Outcome: Mean Change From Baseline on the EORTC QLQ-C30 - Global Heath/QoL
Description: Mean change from baseline on the EORTC QLQ-C30
  The EORTC QLQ-C30 is a 30-item scale composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A higher scale score represents a higher level of well-being and better ability of daily functioning. Thus, a high score for a functional scale represents a high/healthy level of functioning; a high score for the global health status/HRQoL represents a high HRQoL.
Time Frame: At Day 1 and at specific time points up to month 24
Population: PRO Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BB2121
Number analyzed (Participants) | 126
Score on a Scale
  Day 1: number analyzed (Participants) | 114
  Day 1 | -4.7 (17.03)
  Month 1: number analyzed (Participants) | 109
  Month 1 | 4.3 (19.95)
  Month 3: number analyzed (Participants) | 86
  Month 3 | 8.8 (20.31)
  Month 6: number analyzed (Participants) | 76
  Month 6 | 12.5 (19.12)
  Month 9: number analyzed (Participants) | 59
  Month 9 | 15.7 (20.88)
  Month 12: number analyzed (Participants) | 55
  Month 12 | 14.1 (21.57)
  Month 18: number analyzed (Participants) | 26
  Month 18 | 10.6 (17.25)
  Month 24: number analyzed (Participants) | 14
  Month 24 | 7.1 (14.93)

19. Secondary Outcome: Mean Change From Baseline on the EORTC QLQ-MY20 - Disease Symptoms
Description: Mean change from baseline on the EORTC QLQ-MY20
  The EORTC has developed a myeloma module referred to as QLQ- MY20, to be administered alongside the core QLQ-C30. The QLQ-MY20 is a 20-item myeloma module intended for use among patients varying in disease stage and treatment modality.
  All items will be scored from 0 to 100. The average of the scores will represent the symptoms score. A high score for a symptom scale/item represents a high level of symptomatic problem.
Time Frame: At Day 1 and at specific time points up to month 24
Population: PRO Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BB2121
Number analyzed (Participants) | 126
Score on a Scale
  Day 1: number analyzed (Participants) | 114
  Day 1 | -0.8 (14.11)
  Month 1: number analyzed (Participants) | 109
  Month 1 | -10.2 (18.54)
  Month 3: number analyzed (Participants) | 86
  Month 3 | -10.8 (20.32)
  Month 6: number analyzed (Participants) | 75
  Month 6 | -12.6 (20.81)
  Month 9: number analyzed (Participants) | 58
  Month 9 | -14.4 (20.29)
  Month 12: number analyzed (Participants) | 55
  Month 12 | -15.7 (23.28)
  Month 18: number analyzed (Participants) | 26
  Month 18 | -12.0 (20.47)
  Month 24: number analyzed (Participants) | 14
  Month 24 | -13.1 (19.07)

20. Secondary Outcome: Mean Change From Baseline on the EORTC QLQ-MY20 - Side Effects
Description: as for outcome 19
Time Frame: At Day 1 and at specific time points up to month 24
Population: PRO Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BB2121
Number analyzed (Participants) | 126
Score on a Scale
  Day 1: number analyzed (Participants) | 114
  Day 1 | 2.5 (9.51)
  Month 1: number analyzed (Participants) | 109
  Month 1 | 0.0 (11.95)
  Month 3: number analyzed (Participants) | 86
  Month 3 | -2.6 (11.45)
  Month 6: number analyzed (Participants) | 75
  Month 6 | -4.7 (10.16)
  Month 9: number analyzed (Participants) | 58
  Month 9 | -6.5 (10.28)
  Month 12: number analyzed (Participants) | 55
  Month 12 | -4.0 (11.87)
  Month 18: number analyzed (Participants) | 26
  Month 18 | -3.4 (9.96)
  Month 24: number analyzed (Participants) | 14
  Month 24 | -3.2 (7.98)

21. Secondary Outcome: Mean Change From Baseline on the EQ-5D-5L Index
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. The EQ-5D-5L health utility index (HUI) is assessed using the Crosswalk algorithm for France based on the individual responses to the 5 EQ-5D-5L domains ranging from -0.530 to 1.000. The smallest change considered clinically meaningful, is defined as a score difference of 0.08 points.
Time Frame: At Day 1 and at specific time points up to month 24
Population: PRO Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | BB2121
Number analyzed (Participants) | 126
Score on a Scale
  Day 1: number analyzed (Participants) | 115
  Day 1 | 0.0314 (0.1760)
  Month 1: number analyzed (Participants) | 110
  Month 1 | 0.0528 (0.2473)
  Month 3: number analyzed (Participants) | 86
  Month 3 | 0.0998 (0.1956)
  Month 6: number analyzed (Participants) | 76
  Month 6 | 0.0974 (0.1798)
  Month 9: number analyzed (Participants) | 59
  Month 9 | 0.1067 (0.2334)
  Month 12: number analyzed (Participants) | 55
  Month 12 | 0.1097 (0.2287)
  Month 18: number analyzed (Participants) | 26
  Month 18 | 0.1101 (0.2027)
  Month 24: number analyzed (Participants) | 14
  Month 24 | 0.0383 (0.1604)

ADVERSE EVENTS:
Time Frame: From screening to the end of follow up (approximately 5 years and 2 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | BB2121
All-Cause Mortality (participants affected / at risk) | 82/137
Serious Adverse Events (participants affected / at risk) | 108/137
Other Adverse Events (participants affected / at risk) | 137/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BB2121 (N=137)
Anaemia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 12
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 6
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 3
Pericarditis (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Diplopia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 30
Localised oedema (General disorders) | 1
Mucosal inflammation (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 8
Acute graft versus host disease (Immune system disorders) | 1
Cytokine release syndrome (Immune system disorders) | 22
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2
Acute sinusitis (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 2
Coronavirus infection (Infections and infestations) | 1
Device related bacteraemia (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Gastroenteritis salmonella (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Hepatitis E (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Hypopyon (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Listeriosis (Infections and infestations) | 1
Lower respiratory tract infection viral (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 15
Pneumonia aspiration (Infections and infestations) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pneumonia pseudomonal (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 3
Rhinovirus infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 7
Septic shock (Infections and infestations) | 2
Serratia bacteraemia (Infections and infestations) | 1
Typhoid fever (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hyphaema (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Stress fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
C-reactive protein increased (Investigations) | 3
Coronavirus test positive (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Adult failure to thrive (Metabolism and nutrition disorders) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Amnesia (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Cauda equina syndrome (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 2
Cognitive disorder (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Hypotonia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Metabolic encephalopathy (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 4
Delirium (Psychiatric disorders) | 3
Disorientation (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 3
Mood altered (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Chronic kidney disease (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Distributive shock (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Pelvic venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BB2121 (N=137)
Anaemia (Blood and lymphatic system disorders) | 104
Febrile neutropenia (Blood and lymphatic system disorders) | 19
Leukopenia (Blood and lymphatic system disorders) | 70
Lymphopenia (Blood and lymphatic system disorders) | 49
Neutropenia (Blood and lymphatic system disorders) | 130
Thrombocytopenia (Blood and lymphatic system disorders) | 95
Tachycardia (Cardiac disorders) | 22
Constipation (Gastrointestinal disorders) | 45
Diarrhoea (Gastrointestinal disorders) | 61
Dry mouth (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 85
Vomiting (Gastrointestinal disorders) | 34
Asthenia (General disorders) | 22
Chills (General disorders) | 20
Fatigue (General disorders) | 53
Malaise (General disorders) | 7
Oedema peripheral (General disorders) | 27
Pain (General disorders) | 9
Pyrexia (General disorders) | 36
Cytokine release syndrome (Immune system disorders) | 110
Hypogammaglobulinaemia (Immune system disorders) | 32
Candida infection (Infections and infestations) | 8
Influenza (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 10
Pneumonia (Infections and infestations) | 9
Respiratory tract infection (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 21
Urinary tract infection (Infections and infestations) | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 9
Activated partial thromboplastin time prolonged (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 22
Aspartate aminotransferase increased (Investigations) | 26
Blood alkaline phosphatase increased (Investigations) | 18
Blood creatinine increased (Investigations) | 8
C-reactive protein increased (Investigations) | 15
International normalised ratio increased (Investigations) | 7
Weight decreased (Investigations) | 19
Weight increased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 41
Hypercalcaemia (Metabolism and nutrition disorders) | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 15
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 13
Hypoalbuminaemia (Metabolism and nutrition disorders) | 26
Hypocalcaemia (Metabolism and nutrition disorders) | 37
Hypokalaemia (Metabolism and nutrition disorders) | 56
Hypomagnesaemia (Metabolism and nutrition disorders) | 35
Hyponatraemia (Metabolism and nutrition disorders) | 30
Hypophosphataemia (Metabolism and nutrition disorders) | 46
Arthralgia (Musculoskeletal and connective tissue disorders) | 32
Back pain (Musculoskeletal and connective tissue disorders) | 29
Bone pain (Musculoskeletal and connective tissue disorders) | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Dizziness (Nervous system disorders) | 23
Headache (Nervous system disorders) | 47
Somnolence (Nervous system disorders) | 10
Tremor (Nervous system disorders) | 12
Anxiety (Psychiatric disorders) | 19
Confusional state (Psychiatric disorders) | 16
Insomnia (Psychiatric disorders) | 14
Acute kidney injury (Renal and urinary disorders) | 11
Pollakiuria (Renal and urinary disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 12
Hypertension (Vascular disorders) | 19
Hypotension (Vascular disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT03361748/Prot_SAP_000.pdf